CLINICAL TRIAL: NCT05742919
Title: Investigation of Pharmacokinetic Properties of Single Subcutaneous Doses of NNC0194-0499 in Chinese Males
Brief Title: A Research Study Looking at How a Single Dose of the Medicine NNC0194-0499 Behaves in Chinese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9500-4796; U1111-1267-4230 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NNC0194-0499 12 mg (Experimental): Participants will receive a single subcutaneous (s.c.) dose of 12 milligrams (mg) NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499
- NNC0194-0499 30 mg (Experimental): Participants will receive a single s.c. dose of 30 mg NNC0194-0499 on Day 1.
  Interventions: Drug: NNC0194-0499
- NNC0194-0499 96 mg (Experimental): Participants will receive a single s.c. dose of 96 mg NNC0194-0499 on Day 1.
  Interventions: Drug: NC0194-0499

INTERVENTIONS:
Drug: NNC0194-0499 — Participants will receive a single s.c. dose of 12 mg NNC0194-0499 on Day 1.
  Arms: NNC0194-0499 12 mg
Drug: NNC0194-0499 — Participants will receive a single s.c. dose of 30 mg NNC0194-0499 on Day 1.
  Arms: NNC0194-0499 30 mg
Drug: NC0194-0499 — Participants will receive a single s.c. dose of 96 mg NNC0194-0499 on Day 1.
  Arms: NNC0194-0499 96 mg

SUMMARY:
This study looks at how a new study medicine called NNC0194-0499 behaves in the body of Chinese men. Three different dose levels will be tested. Participant will get only one of the three different dose levels of NNC0194-0499. Which dose participant will get will be decided by chance. NNC0194-0499 is a medicine under clinical investigation. It means that the medicine has not yet been approved by the health authorities. Participant will get 1 or 2 injections of the study medicine. It will be injected with a needle into a skin fold on stomach. The study will last for a maximum of 64 days. Participant will not be able to take part in the study if the study doctor considers there is a risk for participant's health.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Chinese male aged 20-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 23.0 and 34.9 kilograms per meter square (kg/m^2) (both inclusive).
* Body weight greater than or equal to 60 kg.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention or related products.
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
AUC0-∞, NNC0194-0499: The area under the NNC0194-0499 serum concentration-time curve from time 0 to infinity after a single dose | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in nanomoles*hours per liter (nmol h/L).

SECONDARY OUTCOMES:
AUC0-168h, NNC0194-0499: The area under the NNC0194-0499 serum concentration-time curve from time 0 to 168 hours after a single dose | From Day 1 (pre-dose) until Day 7 (168 hours)
  Measured in nmol h/L.
Cmax, NNC0194-0499: The maximum concentration of NNC0194- 0499 in serum | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in nmol/L.
tmax, NNC0194-0499: The time from dose administration to maximum serum concentration of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in hours.
t1/2, NNC0194-0499: The terminal half-life of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in hours.
CL/FNNC0194-0499: The apparent total serum clearance of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in liters per hour (L/h).
Vz/FNNC0194-0499: The apparent volume of distribution of NNC0194-0499 in the terminal phase | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in liters (L).
Relative change in triglycerides | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in Percent change.
Relative change in high-density lipoprotein (HDL) cholesterol | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in Percent change.
Relative change in low-density lipoprotein (LDL) cholesterol | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in Percent change.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com